CLINICAL TRIAL: NCT04439344
Title: MATCH Treatment Subprotocol Z1A: Binimetinib in Patients With Tumors (Other Than Melanoma) With NRAS Mutations
Brief Title: Testing Binimetinib as a Potential Targeted Treatment in Cancers With NRAS Genetic Changes (MATCH-Subprotocol Z1A)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-03374; NCI-2020-03374 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAY131-Z1A (Other: ECOG-ACRIN Cancer Research Group); EAY131-Z1A (Other: CTEP); U10CA180820 (NIH); U24CA196172 (NIH)
Record Dates: First submitted 2020-06-18; First posted 2020-06-19 (Actual); Results first posted 2021-08-17 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Advanced Lymphoma; Advanced Malignant Solid Neoplasm; Hematopoietic and Lymphoid Cell Neoplasm; Refractory Lymphoma; Refractory Malignant Solid Neoplasm; Refractory Multiple Myeloma
MeSH Terms: conditions — Hematologic Neoplasms; Lymphoma; Multiple Myeloma | interventions — binimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (binimetinib) (Experimental): Patients receive binimetinib PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Binimetinib

INTERVENTIONS:
Drug: Binimetinib — Given PO
  Other Names: ARRY 162; ARRY 438162; ARRY-162; ARRY-438162; ARRY162; ARRY438162; MEK 162; MEK-162; MEK162; Mektovi

SUMMARY:
This phase II MATCH treatment trial investigates the good and bad effects of binimetinib in patients whose cancer has a genetic change called NRAS mutation. Binimetinib blocks proteins called MEK1 and MEK2, which may be needed for cancer cell growth when an NRAS mutation is present. Researchers hope to learn if binimetinib will shrink this type of cancer or stop its growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the proportion of patients with objective response (OR) to targeted study agent(s) in patients with advanced refractory cancers/lymphomas/multiple myeloma.

SECONDARY OBJECTIVES:

I. To evaluate the proportion of patients alive and progression free at 6 months of treatment with targeted study agent in patients with advanced refractory cancers/lymphomas/multiple myeloma.

II. To evaluate time until death or disease progression. III. To identify potential predictive biomarkers beyond the genomic alteration by which treatment is assigned or resistance mechanisms using additional genomic, ribonucleic acid (RNA), protein and imaging-based assessment platforms.

IV. To assess whether radiomic phenotypes obtained from pre-treatment imaging and changes from pre- through post-therapy imaging can predict objective response and progression free survival and to evaluate the association between pre-treatment radiomic phenotypes and targeted gene mutation patterns of tumor biopsy specimens.

OUTLINE:

Patients receive binimetinib orally (PO) twice daily (BID) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months if less than 2 years from study entry, and then every 6 months for year 3 from study entry.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have met applicable eligibility criteria in the Master MATCH Protocol prior to registration to treatment subprotocol
* Patients must have NRAS mutation in codon 12, 13, 61 as determined via the MATCH Master Protocol
* Patients must have an electrocardiogram (ECG) within 8 weeks prior to treatment assignment and must have no clinically significant abnormalities in rhythm, conduction or morphology of resting ECG (e.g. complete left bundle branch block, third degree heart block)
* Creatinine =< 1.5 mg/dL, or calculated creatinine clearance (determined as per Cockcroft-Gault) >= 50mL/min
* Patients must have adequate cardiac function:

  * Left ventricular ejection fraction (LVEF) >= 50% as determined by a multigated acquisition (MUGA) scan or echocardiogram,
  * QTc interval =< 480 ms

Exclusion Criteria:

* Patients must not have known hypersensitivity to binimetinib or compounds of similar chemical or biologic composition
* Patients with melanoma are excluded
* Patients must not have any active central nervous system (CNS) lesion (i.e., those with radiographically unstable, symptomatic lesions) and/or leptomeningeal metastases

  * NOTE: Patients treated with stereotactic radiotherapy or surgery are eligible if the patient remained without evidence of CNS disease progression >= 3 months. Patients must be off corticosteroid therapy for >= 3 weeks
* Patients must not have a history or current evidence of retinal vein occlusion (RVO) or predisposing factors to RVO (e.g. uncontrolled glaucoma or ocular hypertension, history of hyperviscosity or hypercoagulability syndromes)
* Patients must not have a history of retinal degenerative disease
* Patients must not have a history of Gilbert's syndrome
* Patients must not have uncontrolled arterial hypertension despite medical treatment
* Patients must not have active hepatitis B, and/or active hepatitis C infection
* Patients must not have neuromuscular disorders that are associated with elevated creatine kinase (CK) (e.g., inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy)
* Patients must not have impairment of gastrointestinal function or gastrointestinal disease (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection)
* Patients who have received prior MEK inhibitors are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2016-05-31 (Actual); Primary Completion 2019-05-03 (Actual); Study Completion 2026-03-19 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: James M Cleary, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (1):
- ECOG-ACRIN Cancer Research Group, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subprotocol Z1A was activated on May 31, 2016. A total of 114 patients were assigned to this arm after screening, all from screening cohort. Of the 114 patients, 53 patients were enrolled to arm Z1A in the period from May 31, 2016 and June 7, 2018.
Pre-assignment Details: To be assigned to a specific MATCH subprotocol, patients needed to submit a tumor biopsy for molecular characterization and those with molecular variants addressed by treatments included in the trial entered corresponding MATCH subprotocol. For the subprotocol Z1A, patients had to have a tumor harboring a codon 12, 13, or 61 NRAS-mutation.
Period: Overall Study
Arm/Group | Treatment (Binimetinib)
Started | 53
Started Protocol Therapy | 50
Eligible | 47
Completed (Treatment continued until disease progression or intolerability.) | 0
Not Completed | 53
Not completed — Never started threapy | 3
Not completed — Ineligible | 3
Not completed — Adverse Event | 13
Not completed — Death | 2
Not completed — Disease progression | 29
Not completed — Withdrawal by Subject | 2
Not completed — Alternative therapy | 1

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients
Arm/Group | Treatment (Binimetinib)
Number analyzed (Participants) | 47
Age, Continuous [Median (Full Range); unit: years] | 60 [30 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 40
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 40
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of patients whose tumors have a complete or partial response to treatment among eligible and treated patients. Objective response rate is defined consistent with Response Evaluation Criteria in Solid Tumors version 1.1 criteria for solid tumors, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. For each treatment arm, 90% two-sided binomial exact confidence interval will be calculated for ORR.
Time Frame: Tumor assessments occurred at baseline, then every 2 cycles for the first 26 cycles and every 3 cycles thereafter until disease progression, up to 3 years post registration
Population: Patients who were eligible and received protocol treatment
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Binimetinib)
Number analyzed (Participants) | 47
percentage of participants | 0.021 [0.001 to 0.097]

2. Secondary Outcome: 6-Month Progression-free Survival (PFS) Rate
Description: Progression free survival is defined as time from treatment start date to date of progression or death from any cause, whichever occurs first. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. 6 month PFS rate was estimated using the Kaplan-Meier method, which can provide a point estimate for any specific time point.
Time Frame: Tumor assessments occurred at baseline, then every 2 cycles for the first 26 cycles, and every 3 cycles thereafter until disease progression, up to 3 years post registration, from which 6-month PFS is determined
Population: Patients who were eligible and received protocol treatment
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Binimetinib)
Number analyzed (Participants) | 47
percentage of participants | 0.292 [0.194 to 0.440]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression free survival is defined as time from treatment start date to date of progression or death from any cause, whichever occurs first. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Median PFS was estimated using the Kaplan-Meier method.
Time Frame: Assessed at baseline, then every 2 cycles for the first 26 cycles and every 3 cycles thereafter until disease progression, up to 3 years post registration
Population: Patients who were eligible and received protocol treatment
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Binimetinib)
Number analyzed (Participants) | 47
months | 3.5 [1.8 to 5.8]

ADVERSE EVENTS:
Time Frame: Assessed every 28 days while on treatment and for 30 days after the end of treatment, up to 3 years post registration.
Description: All 53 patients enrolled to the trial were monitored for mortality, the 50 treated patients were monitored for adverse events.
Arm/Group | Treatment (Binimetinib)
All-Cause Mortality (participants affected / at risk) | 43/53
Serious Adverse Events (participants affected / at risk) | 24/50
Other Adverse Events (participants affected / at risk) | 44/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Binimetinib) (N=50)
Heart failure (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Edema limbs (General disorders) | 1
Fatigue (General disorders) | 1
Multi-organ failure (General disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 3
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
CPK increased (Investigations) | 2
Ejection fraction decreased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 2
White blood cell decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1
Syncope (Nervous system disorders) | 1
Eye disorders - Other, specify (Eye disorders) | 1
Hypertension (Vascular disorders) | 6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Binimetinib) (N=50)
Anemia (Blood and lymphatic system disorders) | 7
Edema face (General disorders) | 5
Edema limbs (General disorders) | 17
Fatigue (General disorders) | 18
General disorders and administration site conditions - Other (General disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 8
Rash acneiform (Skin and subcutaneous tissue disorders) | 27
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 4
Constipation (Gastrointestinal disorders) | 6
Diarrhea (Gastrointestinal disorders) | 26
Mucositis oral (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 15
Vomiting (Gastrointestinal disorders) | 9
Alanine aminotransferase increased (Investigations) | 8
Alkaline phosphatase increased (Investigations) | 9
Aspartate aminotransferase increased (Investigations) | 17
CPK increased (Investigations) | 16
Creatinine increased (Investigations) | 4
Lymphocyte count decreased (Investigations) | 4
Neutrophil count decreased (Investigations) | 3
Platelet count decreased (Investigations) | 6
White blood cell decreased (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 5
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 7
Hypocalcemia (Metabolism and nutrition disorders) | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Blurred vision (Eye disorders) | 9
Retinal detachment (Eye disorders) | 3
Eye disorders - Other, specify (Eye disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Hypertension (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol (2018-05-16): https://cdn.clinicaltrials.gov/large-docs/44/NCT04439344/Prot_001.pdf